CLINICAL TRIAL: NCT03323307
Title: Low Cost Optical Coherence Tomography for Point of Care
Brief Title: Low Cost OCT for Point of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Wallace H. Coulter Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00087122
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Optical Coherence Tomography (OCT) of the Retina
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OCT imaging (Experimental): OCT device images retina
  Interventions: Device: OCT imaging

INTERVENTIONS:
Device: OCT imaging — imaging of retina using OCT device

SUMMARY:
The purpose of this study is to compare the performance of a prototype optical coherence tomography (OCT) machine with currently available high resolution OCT machines.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to receive standard OCT testing as part of their clinical visit

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wax, Ph.D., Principal Investigator — Duke University
Locations (1):
- University of North Carolina Kittner Eye Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OCT Imaging: All participants had retinal OCT imaging of both eyes. All participants were first imaged with the commercially available Heidelberg Engineering Spectralis OCT machine. All participants were then imaged with the Low Cost OCT device designed by the study team.
Period: Overall Study
Arm/Group | OCT Imaging
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OCT Imaging
Number analyzed (Participants) | 70
Age, Customized [Count of Participants; unit: Participants]
  <= 50 years | 12
  50 - 59 years | 6
  60 - 69 years | 9
  70 - 79 years | 13
  80 - 89 years | 7
  >= 90 years | 1
  Unknown or Not Reported | 22
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 29
  Female | 40
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 48
  More than one race | 0
  Unknown or Not Reported | 11
Retinal Pathology [Count of Participants; unit: Participants]
  Participants with Retinal Pathology | 38
  Healthy Volunteers | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acceptable OCT Image Quality
Description: measured by: ability to see clearly defined and recognizable structures of the retina with the low cost OCT device
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | OCT Imaging
Number analyzed (Participants) | 70
Participants | 60

2. Secondary Outcome: Central Macular Thickness
Description: compare measurements of central macular thickness obtained with low cost OCT system and Heidelberg Spectralis OCT system
Time Frame: day 1
Population: The current version of the low cost OCT device only acquired a single line image on the retina per scan, which did not allow for the pinpointing of the central macula. Therefore, central macular thickness could not be measured.
Arm/Group | OCT Imaging
Number analyzed (Participants) | 0

3. Secondary Outcome: Total Macular Volume
Description: compare total macular volume measurements obtained with low cost OCT system and Heidelberg Spectralis OCT system
Time Frame: day 1
Population: Volumetric imaging was not achievable with the current version of the low cost OCT device due to the line rate being too slow. Volumetric imaging was possible on the Heidelberg Spectralis OCT, but at a significant increase in acquisition time, which was not feasible for amount of time we had with each subject.
Arm/Group | OCT Imaging
Number analyzed (Participants) | 0

4. Post Hoc Outcome: Contrast-to-Noise Ratio (CNR)
Description: Measure of OCT image quality comparing level of image contrast to level of background noise. CNR = (mean of signal of region of interest [i.e., retina] - mean of background noise) divided by square root of (the square of the standard deviation of the region of interest + the square of the standard deviation of the background noise). Therefore, CNR is unitless.
Time Frame: day 1
Population: Participants from whom OCT images of acceptable quality were obtained.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | OCT Imaging
Number analyzed (Participants) | 60
unitless
  Heidelberg Spectralis OCT device | 1.687 (0.027)
  Low Cost OCT device | 1.592 (0.021)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | OCT Imaging
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

LIMITATIONS AND CAVEATS:
Acquiring data for the secondary endpoints was not feasible given the technical limitations of the current low cost OCT system set up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03323307/Prot_SAP_000.pdf